CLINICAL TRIAL: NCT00353665
Title: Phase 2-3 - Memantine for Disability in Amyotrophic Lateral Sclerosis
Brief Title: Memantine for Disability in Amyotrophic Lateral Sclerosis (MEDALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Mamede de Carvalho, Instituto de Medicina Molecular
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002-04
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; motor neuron disease; memantine; clinical trial
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Memantine; Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - active (Experimental): memantine + riluzole
  Interventions: Drug: Memantine (Ebixa); Drug: riluzole
- 2 (Placebo Comparator): riluzole + placebo
  Interventions: Drug: riluzole; Drug: Placebo

INTERVENTIONS:
Drug: Memantine (Ebixa) — 10 mg bid
  Other Names: Ebixa
  Arms: 1 - active
Drug: riluzole — riluzole 50 mg bid
  Other Names: rilutek
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this trial is to study the effect of Memantine (uncompetitive, moderate affinity, NMDA receptor antagonist that binds to the NMDA receptor channel, and regulates the calcium influx into the neurons), a drug used to treat Alzheimer´s disease, on the progression of Amyotrophic Lateral Sclerosis (ALS). Memantine is added to riluzole (the single drug approved to treat ALS).

DETAILED DESCRIPTION:
Phase 2/3 trial in ALS patients Double-blinded, parallel, randomized (2 blocs, bulbar/spinal onset)

Memantine + riluzole x Placebo + Memantine

Inclusion criteria:

* < 75 years at disease onset
* < 3 years of disease progression
* ALS-FRS > 24
* FVC > 60
* Probable or definite disease (revised El Escorial criteria)
* No other medical condition
* Normal blood tests
* Regular medication on riluzole > 1 month
* Nerve conduction studies ruling out conduction block
* EMG with widespread loss of motor units (revised El Escorial criteria)
* At least one hand with ADM strength > 2 on MRC scale

Duration - 2 years

Evaluation - every 3 months

Primary outcome - ALS-FRS Secondary -SF36, Hamilton depression scale, motor unit number estimation, neurophysiological index, strength (clinical evaluation); side-effects

Intention to treat analysis

60 patients

number estimated for 50% change in decline rate of ALS-FRS

ELIGIBILITY:
Inclusion Criteria:

* Definite or probable disease - revise El Escorial criteria
* Normal blood tests
* Riluzole treatment during 1 month or more
* EMG in accordance with El Escorial criteria

Exclusion Criteria:

* Other diseases (such as PNP)
* Both ADM muscles < 3 on MRC scale
* Conduction block on nerve conduction tests
* Disease duration > 3 years
* ALS-FRS < 25
* Forced vital capacity - <60%

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
ALS-FRS | 12 months

SECONDARY OUTCOMES:
QoL, depression scale, strength (clinical evaluation), forced vital capacity | 12 months
neurophysiology (motor unit counting, neurophysiological index) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mamede de Carvalho, MD, Principal Investigator — Department of Neurology- Hospital de Santa Maria
Locations (1):
- Department of Neurology - Hospital de Santa Maria, Lisbon, Portugal